CLINICAL TRIAL: NCT07116694
Title: Assessment of Acute Psychomotor Agitation Measures Associated With Schizophrenia and Bipolar Disorder
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BioXcel Therapeutics Inc (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BXCL501-402
Record Dates: First submitted 2025-07-07; First posted 2025-08-11 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Bipolar I Disorder; Bipolar II Disorder; Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorders; Psychomotor Agitation
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia; Psychotic Disorders; Psychomotor Agitation | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BXCL501 Sublingual film (Experimental): Experimental: 120 mcg of BXCL501 Sublingual film containing 120 Micrograms Dexmedetomidine
  Interventions: Drug: BXCL501 Sublingual Film

INTERVENTIONS:
Drug: BXCL501 Sublingual Film — Single dose BXCL501 120 mcg
  Other Names: Dexmedetomidine

SUMMARY:
This open-label study will utilize treatment with BXCL501 in order to assess the suitability of patient-and lay informant-assessed outcome measures for evaluation of severity of psychomotor agitation episodes in patients with Bipolar Disorders, Schizophrenia, Schizoaffective, and Schizophreniform disorders and correlate them with clinician-assessed ratings.

DETAILED DESCRIPTION:
This is an open-label study to assess acute psychomotor agitation measures in patient-informant dyads with adult (18-75 years old) males and females experiencing an agitation episode associated with bipolar I disorder, bipolar II disorder, schizophrenia, schizoaffective disorder, or schizophreniform disorder. This validation study will include collecting data from approximately 30 patient-informant dyads during and following an acute psychomotor agitation episode. Data will be collected during the episodes from the dyads and the clinical rater for up to two hours after baseline. The aim of the informant, patient, and investigator ratings will be to assess rater agreement between investigators and informants, as well as investigators and patients.

ELIGIBILITY:
Inclusion Criteria for Participant:

1. Male and female patients 18 to 75 years old, inclusive.
2. Patients who can read, understand, and provide written informed consent.
3. Patients who meet the Diagnostic and Statistical Manual of Mental Disorders, v5, Text Revision (DSM-5-TR) criteria for a primary diagnosis of bipolar I or bipolar II disorder, schizophrenia, schizoaffective or schizophreniform disorder.
4. Patients who, in the opinion of the principal investigator, are in good general health prior to study participation as determined by a detailed medical history, a physical examination, and a 12-lead electrocardiogram (ECG).
5. Female participants, if of child-bearing potential and sexually active, and male participants, if sexually active with a partner of child-bearing potential, agree to use a medically acceptable and effective birth control method throughout the study and for one month following the end of the study.
6. Based on history, in the past 30 days prior to Screening, patients must have had at least one clinical presentation of agitation requiring intervention.
7. Patients who are receiving stable psychotropic treatment for 30 days prior to Screening for the underlying primary diagnosis and who are expected to remain on stable treatment for the duration of the study.

Inclusion Criteria for Informant:

1. At least 18 years of age at the time of screening.
2. Is a spouse, significant other, family member, friend, home health aide, or residence manager of an adult patient who:

   1. Has a clinical diagnosis of bipolar I or bipolar II disorder, schizophrenia, schizoaffective or schizophreniform disorder.
   2. Is determined to be eligible for the study per the patient inclusion/exclusion criteria.
3. Has known the patient for at least 12 months cumulatively.
4. Currently living with or routinely contacting the patient at least five days a week.
5. Does not plan to discontinue contact with the patient during the study period.
6. Willing and able to provide written informed consent.

Exclusion Criteria for Participant:

1. Patients with serious or unstable medical illnesses. These include current hepatic (moderate-severe hepatic impairment), renal, gastroenterological, respiratory, cardiovascular (including ischemic heart disease, congestive heart failure), endocrinologic, or hematologic disease.
2. Psychiatric comorbidities are generally allowed; however, moderate or severe substance use disorders (SUD) (within the past 6 months) are exclusionary if the substance involved is other than nicotine or caffeine.
3. The investigator believes the patient has a history of agitation episodes due to substance use.
4. A diagnosis of antisocial personality disorder, borderline personality disorder, or narcissistic personality disorder that predated the diagnosis of schizophrenia or bipolar disorder, or in the opinion of the Investigator, is independent of the signs and symptoms of the schizophrenia or bipolar disorder.
5. Suicidality as assessed with the Columbia Suicide Severity Rating Scale (C-SSRS). Clinically significant risk of suicide based on the Investigator's clinical opinion or a history of an actual suicide attempt in the last year are also exclusionary.
6. Female patients who have a positive pregnancy test at screening/baseline or are breastfeeding.
7. Currently treated with alpha-1 noradrenergic blockers (terazosin, doxazosin, tamsulosin, alfuzosin, or prazosin), alpha-2 adrenergic agonists, or other prohibited medications.
8. Patients with hydrocephalus, seizure disorder, or history of significant head trauma, stroke, transient ischemic attack, subarachnoid bleeding, brain tumor, encephalopathy, meningitis, Parkinson's disease, or focal neurological findings.
9. Patients with ECG abnormalities considered clinically significant by the Investigator or qualified designee with clinical implications for the patient's participation in the study.
10. Patients who have received an investigational drug within 30 days prior to Baseline.
11. For any reason, patients considered by the Investigator, or designee, to be unsuitable candidates for receiving dexmedetomidine, e.g., patients with a history of allergic reactions to dexmedetomidine.

Exclusion Criteria for Informant:

1. Appears to have an impairment (e.g., cognitive, hearing, visual) or insufficient knowledge of the English language that could interfere with their ability to provide written consent, complete written assessments, or an interview (based on screener judgment).
2. Unable to accompany the patient and remain present at the clinical site to complete ratings for the full two-hour data collection period while the patient experiences an acute agitation episode that needs to be treated.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Informant and Clinician ratings comparison | Before and 2 hours after the intervention
  The aim of the study is to assess the agreement/correlations among different measures so the comment is correct that different units of measure are being assessed. The informant-completed questionnaire (modified clinical global impression of severity for informants (mCGI-S-INF) and the clinical-rater completed questionnaire, Positive and Negative Syndrome Scale - Excited Component (PEC) are the primary outcomes being assessed. The mCGI-S-INF is a single item with a 0 to 3 point scale with higher values indicating more severe agitation. The PEC is a five item questionnaire with 7-point response options, overall scores range from 5 to 35 with higher scores indicating more severe agitation.
Informant training materials assessment | Within 7 days of the intervention
  Assess content validity of the Modified Clinical Global Impression of Severity for Informants (mCGI-S-INF) and informant training materials. The scale being utilized is mCGI-S-INF. There is no score as it is a qualitative assessment and it is being validated to measure patient informant reported outcomes against patient reported outcomes (mCGI-S-PAT) and physician reported outcomes using the Positive and Negative Syndrome Scale - Excited Component (PEC) scale where the highest score indicates the maximum agitation that could be experienced.

SECONDARY OUTCOMES:
Patient and Clinician ratings comparison | Before and 2 hours after the intervention
  The aim of the study is to assess the agreement/correlations among different measures so the comment is correct that different units of measure are being assessed. The patient-completed questionnaire (modified clinical global impression of severity for patients (mCGI-S-P) and the clinical-rater completed questionnaire, Positive and Negative Syndrome Scale - Excited Component (PEC) are the primary outcomes being assessed. The mCGI-S-P is a single item with a 0 to 3 point scale with higher values indicating more severe agitation. The PEC is a five item questionnaire with 7-point response options, overall scores range from 5 to 35 with higher scores indicating more severe agitation.
Patient training materials assessment | Within 7 days of the intervention
  Assess content validity of the Modified Clinical Global Impression of Severity for Patients (mCGI-S-PAT) training materials. The scale being utilized is mCGI-S-PAT. There is no score as it is a qualitative assessment and is being validated to measure patient reported outcomes against physician reported outcomes using the Positive and Negative Syndrome Scale - Excited Component (PEC) scale where the highest score indicates the maximum agitation that could be experienced.
Patients completion of the Modified Clinical Global Impression of Severity for Patients (mCGI-S-PAT) | Before and 2 hours after the intervention
  Evaluate whether patients with acute psychomotor agitation can complete the Modified Clinical Global Impression of Severity for Patients (mCGI-S-PAT) evaluation tool. The mCGI-S-PAT is already in the trial protocol and this protocol so it would be disruptive to rename the item at this point. The measure assesses severity of agitation 'right now' with response options of none, mild, moderate, and severe.

CONTACTS AND LOCATIONS:
Overall Officials: Matt Mandel, MD, Study Chair — BioXcel Therapeutics
Locations (5):
- United States (5):
  - BioXcel Clinical Research Site 103, Chino, California
  - BioXcel Clinical Research Site 105, Oceanside, California
  - BioXcel Clinical Research Site 102, Orange, California
  - BioXcel Clinical Research Site 101, St Louis, Missouri
  - BioXcel Clinical Research Site 106, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: No